CLINICAL TRIAL: NCT07046806
Title: Oral Deucrictibant for the Prophylactic and Acute Treatment in Patients With Bradykinin Mediated Angioedema With Normal C1 Inhibitor (BK-AE-nC1INH)
Brief Title: Oral Deucrictibant for Prophylactic and Acute Treatment in Hereditary Angioedema Patients
Acronym: BK-AE-nC1INH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute for Asthma and Allergy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IAA-PHA-ISR01a
Record Dates: First submitted 2025-05-09; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hereditary Angioedema (HAE); Angioedema; Bradykinin-mediated Angioedema; C1 Inhibitor Deficiency
Keywords: Bradykinin; deucrictibant; HAE; BK-AE-nC1INH; nC1INH; C1 Inhibitor; C4
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Deucrictibant XR tablet, 40 mg, prophylaxis (Experimental): Deucrictibant XR tablet, 40 mg, QD, oral use for 12 weeks
  Interventions: Drug: Deucrictibant XR tablet
- Placebo to deucrictibant XR tablet, 40 mg, prophylaxis (Placebo Comparator): Placebo tablets, 40 mg equivalent, QD, oral use for 12 weeks
  Interventions: Drug: Placebo comparator to XR tablet
- On-demand deucrictibant 20 capsule, oral use (Experimental): Single 20 capsule orally for treatment of on-demand angioedema attack, for up to 16 weeks
  Interventions: Drug: Deucrictibant 20 mg capsule
- Placebo comparator to on-demand deucrictibant 20 capsule, oral use (Placebo Comparator): Placebo capsules for treatment of on-demand angioedema attacks, for up to 16 weeks
  Interventions: Drug: Placebo comparator to 20 mg capsule

INTERVENTIONS:
Drug: Deucrictibant XR tablet — Deucrictibant 40 mg XR tablet for prophylaxis
  Other Names: Deucrictibant XR
  Arms: Deucrictibant XR tablet, 40 mg, prophylaxis
Drug: Placebo comparator to XR tablet — Placebo comparator to deucrictibant 40 mg XR tablet, prophylaxis
  Other Names: Placebo
  Arms: Placebo to deucrictibant XR tablet, 40 mg, prophylaxis
Drug: Deucrictibant 20 mg capsule — Deucrictibant active drug for on-demand treatment of angioedma attacks
  Other Names: Deucrictibant
  Arms: On-demand deucrictibant 20 capsule, oral use
Drug: Placebo comparator to 20 mg capsule — Placebo comparator to Deucrictibant 20 mg capsule for on-demand treatment of angioedema attacks
  Other Names: Placebo
  Arms: Placebo comparator to on-demand deucrictibant 20 capsule, oral use

SUMMARY:
To assess the efficacy of prophylactic treatment with deucrictibant extended release (XR) tablet versus placebo in preventing angioedema attacks, and to also assess the efficacy of deucrictibant soft capsules as on-demand treatment versus placebo in achieving angioedema symptom relief during acute attacks.

DETAILED DESCRIPTION:
Study Design:

The study has 2-parts, studying the efficacy of deucrictibant versus placebo for prophylactic and on-demand treatment of angioedema attacks will be assessed in adult participants with BK-AE-nC1INH. Each part of the study is designed a randomized, double-blind, placebo-controlled cross-over trial. Up to 10 patients to be enrolled.

Deucrictibant has been adopted as the international nonproprietary name (INN) for the active ingredient, previously referred to as PHA121 or PHA-022121. Deucrictibant is under development as an orally administered bradykinin B2 receptor antagonist with potential for both acute therapeutic and prophylactic use in patients with different types of BK-mediated angioedema, including HAE-1/2, HAE with normal C1INH, acquired angioedema due to C1INH deficiency, and non-hereditary BK-mediated angioedema with normal C1INH.

Throughout the study (Parts 1 and 2), a diary will be used to record all symptoms and details of angioedema attacks, including on-demand treatments, as well as Patient Reported Outcomes (PROs). Participants need to have access to FDA approved on-demand angioedema medication and be able to treat any angioedema attack that may occur using standard of care on-demand therapies. In addition to the collected data on angioedema attacks, the diary will be used as a dosing diary for the daily intake of study drug treatment in Part 1.

Part 1 will evaluate the efficacy and safety of deucrictibant administered orally for prophylaxis against angioedema attacks in patients with BK-AE-nC1INH. After providing written informed consent, participants will be screened for eligibility. Eligible participants will be enrolled in the study. Participants receiving angioedema medications for long-term prophylaxis (LTP) will discontinue and washout these medications prior to Screening.

Dosing schedule: QD administration of study drug or placebo (double blind) throughout the Treatment Period consisting of deucrictibant (40 mg strength) XR tablet and matching placebo for oral use.

The duration of an individual's participation in Part 1 is up to 24 weeks (12 weeks on each deucrictibant and placebo, in random order).

Participants will be randomized in a 1:1 ratio to receive deucrictibant 40 mg XR tablet or matching placebo once daily (QD) each for 12 weeks and then participants will be crossed over, for a total of 24 weeks of treatment.

Part 2: After completion of Part 1, a study visit will be conducted at Week 24, at which the enrolled participants will be re-randomized in Part 2 on a 1:1 ratio to a treatment sequence to receive deucrictibant 20 mg soft capsule following by matching placebo or vice versa, with one capsule given for each of 2 attacks. Participants will self-administer blinded study drug in the assigned treatment sequence at home to treat 2 non-laryngeal qualifying angioedema attacks (at least one attack symptom [skin pain, skin swelling, or abdominal pain] has reached the individual item score of ≥20 in VAS-3). The time of administration of study drug as well as rescue medication must be recorded in the patient diary.The expected duration of Part 2 is up to 16 weeks.

End-of-Treatment and End-of-Study visits will occur within 7±2 days and 28 days (-14 days), respectively, after treatment of the second attack in Part 2.

Dosing schedule: Administration of study drug for acute angioedema attacks, dosing consists of deucrictibant (20 mg strength) soft capsule and matching placebo for oral use.

The duration of treatment in Part 2 is approximately 16 weeks.

Efficacy will be assessed based upon the occurrences of angioedema attacks, which will be confirmed by Investigators. During Screening, site personnel will discuss with participants the requirements for reporting angioedema attacks, including the information that is to be captured for each angioedema attack.

A Statistical Analysis Plan (SAP) will be finalized prior to database lock and will include a more technical and detailed description of all planned statistical analyses of all study endpoints.

The analysis of safety and tolerability will be performed on the Safety Analysis Set (ie, all randomized participants who have received at least 1 dose of study drug). Treatment-emergent AEs (TEAEs) are defined as AEs that start or pre-existing AEs that have worsened after the initiation of study drug.

The number and percentage of participants with TEAEs will be summarized by treatment group by body system organ class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA®). Clinical laboratory data, vital signs, physical examination, and ECG data will be presented in summary tables and individual listings by treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Male or female, aged ≥18 at the time of provision of informed consent.
3. Diagnosis of bradykinin-mediated angioedema based upon all of the following:

   * Clinical history consistent with angioedema (subcutaneous or mucosal, nonpruritic swelling without accompanying urticaria), not responsive to treatments of anti-histamine, corticosteroid, and/or omalizumab.
   * Tried and failed at least 2 weeks of cetirizine 20 mg twice a day (or its equivalent alternative antihistamines, such as fexofenadine, loratadine, desloratadine or levocetirizine, etc.).
   * Total blood BK peptide levels following 3 days cold activation is above the diagnostic value in non-attack and/or attack period*.

     *The "attack period" is defined as within 24 hours after an attack.
   * Documented diagnostic testing results: C1INH antigen concentration and functional activity within normal range; C4 antigen concentration within normal range.
4. Documented history of at least 2 angioedema attacks in the previous 2 months.
5. Reliable access and experience to use standard of care medication to effectively manage acute angioedema attacks.

Exclusion Criteria:

1. Any diagnosis of angioedema other than BK-AE-nC1INH.
2. Participation in a clinical study with any other investigational drug within the previous 30 days or within 5 half-lives of the investigational drug at Screening (whichever was longer).
3. Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks of Screening.
4. Receiving prophylactic treatment for BK-AE-nC1INH. Participants who have previously received prophylactic therapy but have stopped can participate in this study provided a sufficiently long washout period (≥5 half-life) is observed before the participant is screened. Exclusion includes use of:

   • Short-term prophylaxis for BK-AE-nC1INH within 7 days prior to Screening.
5. Any females who are pregnant, plan to become pregnant, or are currently breast-feeding.
6. Abnormal hepatic function (aspartate aminotransferase >2× upper limit of normal, alanine aminotransferase >2× ULN, or total bilirubin >1.5× upper limit of normal). Participants with Gilbert's syndrome, defined as isolated increase of total bilirubin ≤3× upper limit of normal and aspartate aminotransferase and alanine aminotransferase within the normal range, are not excluded.
7. Abnormal renal function (estimated glomerular filtration rate [eGFR] <60 mL/min/1.73 m2).
8. Any clinically significant history of angina, myocardial infarction, syncope, stroke, left ventricular hypertrophy or cardiomyopathy, uncontrolled hypertension, bradycardia, or any other clinically significant cardiovascular abnormality within the previous year that, in the opinion of the Investigator, would interfere with the participant's safety or ability to participate in the study.
9. History of epilepsy and other significant neurological diseases.
10. Any clinically significant gastrointestinal dysfunction (eg, diarrhea, inflammatory bowel disease) which may impact on study drug absorption.
11. History of alcohol or drug abuse within the previous year, or current evidence of substance dependence or abuse.
12. Use of concomitant medications with systemic absorption that are moderate and strong inhibitors or strong inducers of CYP3A4, such as clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, and grapefruit juice as well as carbamazepine, and rifampin within the last 30◦days or within 5◦half-lives (whichever is longer) of the time of randomization.
13. Known hypersensitivity to deucrictibant or any of the excipients of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Part-1: Incidence and quality of HAE attacks comparing active versus placebo arms. | 24 weeks
  Part-1: Time-normalized number of Investigator-confirmed moderate or severe angioedema attacks during the Treatment Period. Time-normalized number of Investigator-confirmed angioedema attacks treated with on-demand medication during the Treatment Period.
Part-2: Efficacy of active on-demand treatment versus placebo in achieving angioedema symptom relief during acute attacks | 16 weeks
  Part-2: Time to onset of symptom relief of active drug versus placebo, defined as Patient Global Impression of Change (PGI-C) rating of at least "a little better" for 2 consecutive timepoints within 12 hours post-treatment. Time to complete symptom resolution, defined as achieving PGI-S rating of "none" within 48 hours post-treatment.

SECONDARY OUTCOMES:
Safety assessment of oral deucrictibant extended release (XR) tablet (Part 1), and deucrictibant oral on-demand tablets (Part 2). | 40 weeks
  Adverse event severity, expectedness, and relatedness of the active drug, classified based on their severity, whether they were expected, and their potential relationship to the study intervention (Parts 1 and 2).
Part-1: Change in Health-Related Quality of Life (HRQoL) Scores Between Active Drug and Placebo Periods | 16 weeks
  Assessment of quality of life will be conducted using a validated disease-specific instrument, such as the Hereditary Angioedema Quality of Life Questionnaire (HAE-QoL), and supplemented by a daily patient diary Daily diary entries will record the presence or absence of attacks, their severity, duration, body location, treatment used, time to resolution, and the impact on daily living (missed work/school, physical limitations, mood, and social activities).documenting physical, emotional, and functional impacts of each attack.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute For Asthma & Allergy, Wheaton, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial Individual Participant Data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA) at least 9 months after the publication date.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 9 months post publication date of the clinical trial data.
Access Criteria: Any qualified researchers engaging in independent scientific research.

REFERENCES:
- [Background] Weller K, Groffik A, Magerl M, Tohme N, Martus P, Krause K, Metz M, Staubach P, Maurer M. Development and construct validation of the angioedema quality of life questionnaire. Allergy. 2012 Oct;67(10):1289-98. doi: 10.1111/all.12007. Epub 2012 Aug 23. PMID 22913638
- [Background] Riedl MA, Danese M, Danese S, Ulloa J, Maetzel A, Audhya PK. Hereditary Angioedema With Normal C1 Inhibitor: US Survey of Prevalence and Provider Practice Patterns. J Allergy Clin Immunol Pract. 2023 Aug;11(8):2450-2456.e6. doi: 10.1016/j.jaip.2023.01.023. Epub 2023 Jan 30. PMID 36720386
- [Background] Lumry WR, Li HH, Levy RJ, Potter PC, Farkas H, Moldovan D, Riedl M, Li H, Craig T, Bloom BJ, Reshef A. Randomized placebo-controlled trial of the bradykinin B(2) receptor antagonist icatibant for the treatment of acute attacks of hereditary angioedema: the FAST-3 trial. Ann Allergy Asthma Immunol. 2011 Dec;107(6):529-37. doi: 10.1016/j.anai.2011.08.015. Epub 2011 Oct 5. PMID 22123383